CLINICAL TRIAL: NCT03377686
Title: The Feasibility and Diagnostic Value of New Point-of-care Instruments for Breath Analysis in Children With Asthma, Cystic Fibrosis (CF), and Healthy Controls
Brief Title: Breath Analysis in Children by New Point-of-care Instruments
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL 53995.068.15
Record Dates: First submitted 2016-01-29; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Asthma; Cystic Fibrosis
Keywords: paediatrics; breath analysis; volatile organic compounds; respiratory diseases
MeSH Terms: conditions — Asthma; Cystic Fibrosis; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — inflammation markers in exhaled breath
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asthma: Inflammation markers in exhaled breath will be used in 20 children aged 6 to 16 years with doctor's diagnosed asthma
  Interventions: Diagnostic Test: inflammation markers in exhaled breath
- Cystic fibrosis: Inflammation markers in exhaled breath will be used in 20 children aged 6 to 16 years with CF
  Interventions: Diagnostic Test: inflammation markers in exhaled breath
- Healthy: Inflammation markers in exhaled breath will be used in 20 children aged 6 to 16 years old without respiratory diseases
  Interventions: Diagnostic Test: inflammation markers in exhaled breath

INTERVENTIONS:
Diagnostic Test: inflammation markers in exhaled breath — non-invasive, cross-sectional, assessment of inflammation markers in exhaled breath with various techniques (observational)

SUMMARY:
In this study new hand-held devices for measuring exhaled breath will be tested in children with asthma, CF, and healthy controls. Main objectives will be feasibility and discriminative value of these techniques.

DETAILED DESCRIPTION:
Rationale: Assessment of volatile organic compounds (VOCs) is a new recently developed non-invasive technique to assess airway inflammation. The non-invasive character makes it highly suitable for use in (preschool) children. However, the analysis of VOCs by gas chromatography mass spectrometry technique (GC-MS), the gold standard, is expensive and time consuming. Therefore, new hand-held devices (such as electronic Noses (eNoses) and Ion Mobility Spectrometer techniques) have been developed. However, these new point-of-care instruments have not been studied in children.

Objectives: 1) To test whether new point-of-care instruments for the measurement of VOCs in exhaled breath are feasible for use in children aged 6 to 16 years; 2) To explore whether these techniques can differentiate between healthy children, asthmatic children and children with Cystic Fibrosis (CF).

Study design: Cross-sectional study design. Several VOCs tests will be performed in all participants.Besides, fraction of exhaled nitric oxide (FeNO) and inflammatory markers in exhaled breath condensate (EBC) will be measured.

Study population: Three groups of children aged 6 to 16 years: 20 healthy children, 20 children with doctor's diagnosed asthma, 20 children with CF.

Main study parameters/endpoints: Each technique will be evaluated for its use and feasibility in children. For each technique, VOC profiles between study groups will be evaluated for its discriminative power.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 16 years
* Healthy group: See exclusion criteria
* Asthma group: Doctor's diagnosed asthma
* Cystic Fibrosis group: A diagnosis of cystic fibrosis, confirmed by a sweat test or genetic analysis

Exclusion criteria

* Recent course of prednisone or antibiotics (< 1 month before test)
* Passive smoking
* Other chronic inflammatory disease (e.g. inflammatory bowel disease, rheumatic disease, auto-immune disease)
* Healthy children:

  * No current or history of respiratory symptoms
  * No current or history of allergic rhinitis

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Three groups of children aged 6 to 16 years: 20 healthy children, 20 children with doctor's diagnosed asthma, 20 children with CF.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events directly related to the various point-of-care tests used | Questionnaire will be done directly after specific test (1 day). No long term (S)AE is expected and measurement of each test is only performed once.
  Any adverse event of any kind will be noted. Furthermore, each participant will be asked whether the test was easy to perform. This question can be answered on a 5-point scale (0=totally agree that test was easy to perform, 4= totally disagree that test was easy to perform)

SECONDARY OUTCOMES:
Sensitivity and Specificity of new point-of-care Aeonose eNose in diagnosing asthma. | Measurements will be analysed within 6 to 12 months
  Aeonose eNose measurements will be analysed by in house software program (Aethena) developed by eNose company (Zutphen, Netherlands). To test sensitivity and specificity, first an area under the receiver operating curve must be calculated with the aforementioned software program. Hereafter sensitivity and specificity of the eNose can be calculated.
Sensitivity and Specificity of new point-of-care Aeonose eNose in diagnosing cystic fibrosis. | Measurements will be analysed within 6 to 12 months
  Aeonose eNose measurements will be analysed by in house software program (Aethena) developed by eNose company (Zutphen, Netherlands). To test sensitivity and specificity, first an area under the receiver operating curve must be calculated with the aforementioned software program. Hereafter sensitivity and specificity of the eNose can be calculated.
Sensitivity and Specificity of Ion Mobility Spectrometry in diagnosing asthma. | Measurements will be analysed within 6 to 12 months
  IMS measurements will be analysed by software program developed for using IMS data (Visual Now, Ganshorn, Dortmund, Germany). By IMS different VOCs peaks are generated. By using the aforementioned software, these peaks can be analysed and sensitivity and specificity between asthma and healthy children can be calculated.
Sensitivity and Specificity of Ion Mobility Spectrometry in diagnosing cystic fibrosis. | Measurements will be analysed within 6 to 12 months
  IMS measurements will be analysed by software program developed for using IMS data (Visual Now, Ganshorn, Dortmund, Germany). By IMS different VOCs peaks are generated. By using the aforementioned software, these peaks can be analysed and sensitivity and specificity between CF and healthy children can be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Dompeling, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bannier MAGE, van de Kant KDG, Jobsis Q, Dompeling E. Feasibility and diagnostic accuracy of an electronic nose in children with asthma and cystic fibrosis. J Breath Res. 2019 May 8;13(3):036009. doi: 10.1088/1752-7163/aae158. PMID 30213921